CLINICAL TRIAL: NCT07378319
Title: Effectiveness of Ultrasound-Guided Dextrose Prolotherapy for Persistent Chest Wall and Axillary Symptoms in Breast Cancer Survivors: A Prospective Case Series.
Brief Title: Dextrose Prolotherapy for Post-Breast Cancer Chest Wall and Axillary Tightness.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGHTHU114122
Record Dates: First submitted 2026-01-15; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Females
Keywords: breast cancer; dextrose injection
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study utilizes a prospective, single-arm, interventional model (Single Group Assignment) designed as a pilot case series. The design focuses on evaluating the within-subject changes in functional and pain-related outcomes following a standardized interventional protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Participants in this single experimental arm will receive three sessions of ultrasound-guided dextrose injections (e.g., 5% or 15% Dextrose) targeting symptomatic myofascial and interfascial planes of the ipsilateral chest wall and axilla, such as the pectoralis major-minor interface or axillary fascia. Injections are administered at 4-week intervals (at Baseline, Week 4, and Week 8). Throughout the 6-month study period, all participants continue their standardized rehabilitation program, which includes range-of-motion exercises, stretching of the chest wall and axillary musculature, and progressive strengthening.
  Interventions: Procedure: ultrasound guided dextrose prolotherapy

INTERVENTIONS:
Procedure: ultrasound guided dextrose prolotherapy — Participants receive three sessions of ultrasound-guided 5% dextrose injections into symptomatic myofascial and interfascial planes of the ipsilateral chest wall and axillary region. The technique involves identifying areas of soft-tissue thickening or restricted fascial glide under high-frequency ultrasound. Injection targets are individualized to each patient's specific site of restriction (e.g., clavipectoral fascia, pectoralis major-minor interface, or axillary fascia). Sessions are administered at 4-week intervals (at weeks 0, 4, and 8).

SUMMARY:
The goal of this clinical trial (prospective case series) is to evaluate the feasibility, safety, and preliminary clinical outcomes of ultrasound-guided dextrose prolotherapy in female breast cancer survivors with persistent ipsilateral chest wall and axillary pain and tightness who have plateaued with standard physical therapy.

The main questions it aims to answer are:

Does ultrasound-guided dextrose prolotherapy significantly improve upper extremity functional limitation (measured by the QuickDASH questionnaire)?

What are the effects of this intervention on pain intensity (NRS), active shoulder range of motion (AROM), and anterior chest wall soft-tissue tightness (pectoralis minor muscle length)?

Participants will:

Undergo a comprehensive baseline physical examination and ultrasound assessment of the symptomatic chest wall and axilla.

Receive three sessions of ultrasound-guided 5% dextrose injections into targeted soft-tissue planes at 4-week intervals.

Continue their designated standard rehabilitation program, including range-of-motion and stretching exercises.

Attend follow-up assessments at 4-week intervals during the treatment phase, with long-term follow-up at 3 and 6 months after the final injection to evaluate the durability of the response.

DETAILED DESCRIPTION:
Detailed Description Post-surgical breast cancer survivors often experience persistent shoulder and upper-quarter dysfunction characterized by chest wall and axillary tightness. While conventional physical therapy focuses on joint mobilization and stretching, a subset of patients with significant soft-tissue fibrosis and scar adhesions-patterns reflecting extra-articular restriction-remains non-responsive to standard care.

This prospective case series evaluates the role of ultrasound-guided dextrose prolotherapy as a targeted intervention for this challenging clinical problem. The rationale is based on the mechanical and biological effects of dextrose-based hydrodissection, which aims to separate adherent fascial planes and promote tissue remodeling in areas of postoperative myofascial restriction.

Procedural Workflow:

Scanning Protocol: A high-frequency linear transducer is used to systematically scan the ipsilateral pectoral and axillary regions. The physician identifies symptomatic areas characterized by tissue thickening, loss of normal fascial glide, or focal tenderness.

Injection Technique: Using a sterile, ultrasound-guided approach, a dextrose solution is administered into the identified myofascial or perimysial planes. The injection targets are individualized based on each participant's specific site of restriction (e.g., between the pectoralis major and minor muscles or within the axillary fascia).

Frequency and Duration: Participants receive a total of three injection sessions spaced 4 weeks apart. This interval allows for the observation of cumulative clinical effects and soft-tissue adaptation.

Integrated Care: To maximize functional gains, all participants continue a standardized, home-based rehabilitation program consisting of progressive stretching and postural correction throughout the 6-month study period.

The study aims to provide preliminary data on whether this interventional approach can bridge the therapeutic gap for survivors with persistent myofascial symptoms despite prior rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* History of breast cancer surgery (mastectomy or breast-conserving surgery), with or without axillary lymph node dissection
* Persistent ipsilateral chest wall and/or axillary pain, tightness, or movement restriction lasting ≥ 3 months after surgery;
* Clinically significant baseline symptom severity, defined as Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire ≥ 25 and/or pain intensity ≥ 5/10 on the Numeric Rating Scale (NRS);
* Completion of 12 weeks of standard physical therapy with no significant improvement, defined as a change in QuickDASH score from baseline to completion of therapy below the minimal clinically important difference (MCID; <15 points ) and/or pain improvement < 2 points on the NRS .
* Age ≥ 18 years;
* Ability to provide written informed consent.

Exclusion Criteria:

* Evidence of local cancer recurrence or metastatic disease;
* Active lymphedema requiring ongoing decongestive therapy at the time of enrollment;
* Shoulder pathology, including intra-articular or peri-articular conditions (e.g., adhesive capsulitis with marked capsular restriction, or acute rotator cuff tear,) judged by clinical assessment to be the dominant cause of symptoms.
* Active infection, skin lesion, or unhealed surgical wound at the intended injection site;
* Known bleeding disorders or anticoagulant use contraindicating injection;
* Known allergy to dextrose or any components of the injection protocol;
* Pregnancy or other medical conditions precluding participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-11 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Upper Extremity Function | Baseline, 4 weeks after the 1st injection, 4 weeks after the 2nd injection, 4 weeks after the 3rd injection (approx. 12 weeks from baseline), 3 months after the 3rd injection and 6 months after the 3rd injection
  Upper extremity functional limitation was assessed using the QuickDASH questionnaire, with scores ranging from 0 (no disability) to 100 (most severe disability). The minimal clinically important difference (MCID) for the QuickDASH was defined as 15 points

SECONDARY OUTCOMES:
Pain Intensity | Baseline, 4 weeks after the 1st injection, 4 weeks after the 2nd injection, 4 weeks after the 3rd injection (approx. 12 weeks from baseline), 3 months after the 3rd injection and 6 months after the 3rd injection
  Pain intensity was measured using the Numeric Rating Scale (NRS), with scores ranging from 0 (no pain) to 10 (worst imaginable pain). Participants were instructed to rate their pain intensity during provoked overhead activity or movements that most reliably reproduced their symptoms. A change of ≥ 2 points on the NRS was considered clinically meaningful
Shoulder Range of Motion | Baseline, 4 weeks after the 1st injection, 4 weeks after the 2nd injection, 4 weeks after the 3rd injection (approx. 12 weeks from baseline), 3 months after the 3rd injection and 6 months after the 3rd injection
  Active shoulder range of motion (AROM) was measured using a standard goniometer, including forward flexion and abduction, the most consistently assessed directions across prior studies
Pectoralis Minor Length | Baseline, 4 weeks after the 1st injection, 4 weeks after the 2nd injection, 4 weeks after the 3rd injection (approx. 12 weeks from baseline), 3 months after the 3rd injection , and 6 months after the 3rd injection
  Anterior chest wall soft-tissue tightness was assessed by measuring pectoralis minor muscle length. Specifically, the linear distance between the coracoid process and the anterior inferior edge of the fourth rib was measured in the supine position

OTHER OUTCOMES:
Patient Global Impression of Change | 4 weeks after the 1st injection, 4 weeks after the 2nd injection, 4 weeks after the 3rd injection (approx. 12 weeks from baseline), 3 months after the 3rd injection and 6 months after the 3rd injection
  Overall perceived improvement was evaluated using the Patient Global Impression of Change (PGIC) scale. Participants rated their overall change in symptoms since the intervention on a 7-point Likert scale, ranging from 1 (very much worse) to 7 (very much improved). Scores ≧ 5 (minimal improvement) were considered clinically relevant global improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Yuchun Lee, M.D., Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans Genetal Hospital, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in this article (text, tables, figures, and appendices) will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning 6 months and ending 3 years following article publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal. Proposals should be directed to the corresponding author. To gain access, data requestors will need to sign a data access agreement.